CLINICAL TRIAL: NCT03682848
Title: An Open-label, Single Arm Study to Evaluate the Week 48 Efficacy and Safety of a Two-drug Regimen of Dolutegravir/Lamivudine (DTG/3TC) as a Fixed Dose Combination (FDC), in Antiretroviral Therapy (ART)-Naive HIV-1-infected Adolescents, ≥12 to <18 Years of Age Who Weigh at Least 25 kg
Brief Title: Safety and Efficacy of Dolutegravir/Lamivudine (DTG/3TC) in Therapy-naive Human Immunodeficiency Virus-1 (HIV-1) Infected Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 205861
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Results first posted 2022-08-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: HIV Infections
Keywords: Viral load; Dolutegravir; Lamivudine; HIV-1; Fixed dose combination; DOVATO
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir

STUDY DESIGN:
Intervention Model Description: All participants received FDC of DTG/3TC (50/300 mg) once daily.
Masking Description: This was an open-label study hence, there was no masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DTG/3TC FDC (Experimental): Participants received dolutegravir/lamivudine (DTG/3TC) (50/300 mg) Fixed Dose Combination (FDC) tablets orally once daily.
  Interventions: Drug: DTG + 3TC FDC

INTERVENTIONS:
Drug: DTG + 3TC FDC — DTG + 3TC FDC was available as a 50/300 mg tablet to be given orally once daily.

SUMMARY:
First-line antiretroviral regimens are highly efficacious and generally well tolerated. However, as these regimens need to be taken life-long, there is growing concern about long-term toxicities associated with these regimens. Thus, there is great interest from participants and clinicians in unique regimens that might avoid such toxicities by minimizing the number of antiretrovirals without sacrificing long-term antiviral efficacy. DTG plus 3TC is a novel, well-tolerated first-line regimen for HIV-infected treatment- naive participants, limiting the risk of many common adverse reactions associated with other antiretroviral drugs. This study was designed to evaluate the efficacy and safety of DTG/3TC as an FDC in ART-naive HIV-1-infected adolescents who weighed at least 25 kilograms (kg).

The study consisted of a Screening Phase (up to 28 days prior to the first dose of drug), followed by a Treatment Phase (up to 48 weeks). Participants who successfully completed 48 weeks of therapy and continued to receive benefit from DTG/3TC FDC were eligible to enter a 96-week Extension Phase. Study participants who successfully completed both the Treatment Phase through 48 weeks and the Extension Phase through 144 weeks and continued to receive benefit from this two-drug regimen were to continue receiving DTG/3TC FDC in a Continuation Phase (after Week 144) until DTG and 3TC were both locally approved for use as part of a dual regimen and the single entities of DTG and 3TC were available to participants (e.g., through public health services), or the DTG/3TC FDC tablet, if required by local regulations, was locally approved and available (e.g., commercially or through public health services), or the participant no longer derived clinical benefit, or the participant met a protocol-defined reason for discontinuation.

All participants received the FDC of DTG/3TC (50/300 milligrams) once daily.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1-infected adolescents were 12 to <18 years of age at the time of signing the informed consent form.
* Weight was >25 kg at the time of signing the informed consent form.
* Screening plasma HIV-1 RNA was between 1,000 and =500,000 c/mL.
* Participants were antiretroviral-naive (defined as having had no prior therapy with any antiretroviral agent for the treatment of HIV following a diagnosis of HIV-1 infection). Participants who had received ART for prevention of mother-to-child transmission of HIV in the first 3 months of life were allowed. Participants who had received HIV post-exposure prophylaxis (PEP) or pre-exposure prophylaxis (PrEP) in the past were allowed as long as the last PEP/PrEP dose was = 6 months before HIV diagnosis or there was documented HIV seronegativity at least 2 months after the last prophylactic dose and prior to the date of HIV diagnosis.
* Male and female participants were included. A female participant was eligible to participate if she was not pregnant (as confirmed by a negative serum human chorionic gonadotropin [hCG] test at Screening and a negative urine hCG test before Enrollment) and not lactating. Female participants of child-bearing potential who were engaging in sexual activity that could have led to pregnancy had to agree to use one birth-control method from 28 days prior to the first dose of study medication until 4 weeks after the last dose of study medication (and completion of the follow-up visit). Condoms were additionally recommended, as appropriate use was the only contraceptive method effective in preventing HIV-1 transmission. The investigator was responsible for ensuring that participants understood how to properly use these contraceptive methods. All participants in the study were also counseled on safer sexual practices, including the use and benefit/risk of effective barrier methods (e.g., male condoms), as well as on the risk of HIV transmission to an uninfected partner.
* The participant's parent(s) or legal guardian, or the participant, was capable of giving signed informed consent.

Exclusion Criteria:

* Females who were breastfeeding or who planned to become pregnant or breastfeed during the study were excluded.
* Any evidence of active Centers for Disease Control and Prevention (CDC) Stage 3 and/or Category C or World Health Organization (WHO) Stage 4 disease-except cutaneous Kaposi's sarcoma not requiring systemic therapy-and historical or current CD4 cell counts <200 cells/mm³ or CD4 percent <15 percent resulted in exclusion.
* Participants with severe hepatic impairment (Class C) as determined by the Child-Pugh classification were excluded.
* Participants with unstable liver disease (defined by ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, or known biliary abnormalities (except Gilbert's syndrome or asymptomatic gallstones) were excluded.
* Evidence of hepatitis B virus (HBV) infection at Screening led to exclusion as follows: participants positive for HBsAg were excluded; participants negative for anti-HBs but positive for anti-HBc (negative HBsAg) and positive for HBV DNA were excluded. Participants positive for anti-HBc (negative HBsAg) and anti-HBs (past and/or current evidence) were immune to HBV and were not excluded.
* Participants with an anticipated need for any HCV therapy during the first 48 weeks of the study-and for any HCV therapy based on interferon or drugs with potential adverse drug-drug interactions with study treatment throughout the entire study period-were excluded.
* Untreated syphilis infection (positive rapid plasma reagin [RPR] at Screening without clear documentation of treatment) resulted in exclusion. Participants who were at least 24 hours post-completed treatment were eligible.
* Participants with a history of sensitivity to any study medication or its components, or to drugs of the same class, or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicated participation, were excluded.
* Participants with ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, resected non-invasive cutaneous squamous cell carcinoma, or cervical, anal, or penile intraepithelial neoplasia were excluded. Other localized malignancies required agreement between the investigator and Study Medical Monitor for inclusion.
* Participants who, in the investigator's judgment, posed a significant suicide risk were excluded. A recent history of suicidal behavior and/or suicidal ideation could have been considered evidence of serious suicide risk.
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening resulted in exclusion.
* Treatment with radiation therapy, cytotoxic chemotherapeutic agents, or any systemic immune suppressant within 28 days of Screening resulted in exclusion.
* Treatment with any agent with documented activity against HIV-1 in vitro within 28 days of the first study dose resulted in exclusion.
* Receipt of any prohibited medication, and inability or unwillingness to switch to an alternative medication, resulted in exclusion.
* Exposure to an experimental drug or vaccine within 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent (whichever was longer) prior to the first study dose resulted in exclusion.
* Any evidence of pre-existing viral resistance based on any major resistance-associated mutation in Screening or historical results led to exclusion.
* Any verified Grade 4 laboratory abnormality led to exclusion. A single repeat test during Screening was allowed to verify results.
* Any acute laboratory abnormality at Screening that, in the Investigator's opinion, would have precluded participation in the study of an investigational compound resulted in exclusion.
* ALT >5× the upper limit of normal (ULN), or ALT >5× ULN with bilirubin >1.5× ULN (with >35 percent direct bilirubin), resulted in exclusion.
* Creatinine clearance <50 mL/min/1.73 m² using the Schwartz equation resulted in exclusion.
* Children who were wards of the state or government were excluded.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2025-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (7):
- Kenya (2):
  - GSK Investigational Site, Kericho
  - GSK Investigational Site, Kisumu
- South Africa (3):
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Johannesburg
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
Study sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf

REFERENCES:
- [Derived] Puthanakit T, Aurpibul L, Lopez M, Wang M, Ciuffa M, Bontempo G, Cheung SYA, Deprez I, Buchanan AM, Vavro C, McKenna M, Min S, Tan LK. Efficacy and Safety of the Two-Drug Regimen Dolutegravir-Lamivudine in Adolescents Living With HIV-1 Naive to Antiretroviral Therapy at 48 Weeks (DANCE): A Single-Arm, Open-Label, Phase 3b Trial. J Acquir Immune Defic Syndr. 2025 Jun 1;99(2):202-210. doi: 10.1097/QAI.0000000000003655. PMID 39988749

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DTG/3TC FDC
Started | 32
Completed | 20
Not Completed | 12
Not completed — Withdrawal by Subject | 3
Not completed — Site closed | 5
Not completed — Protocol Deviation | 1
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 16.0 (1.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 13
  Asian - South East Asian Heritage | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) Less Than 50 Copies Per Milliliter (c/mL) at Week 48
Description: Percentage of participants with plasma HIV-1 RNA <50 c/mL was assessed at Week 48 according to the Food and Drug Administration (FDA) snapshot algorithm.
Time Frame: Week 48
Population: Intent To Treat-Exposed (ITT-E) population includes all enrolled participants who received at least one dose of DTG/3TC.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Percentage of Participants | 81 [64 to 93]

2. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <200 c/mL at Week 24
Description: Percentage of participants with plasma HIV-1 RNA <200 c/mL was assessed at Week 24 according to the FDA snapshot algorithm.
Time Frame: Week 24
Population: Intent To Treat-Exposed
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Percentage of Participants | 91 [75 to 98]

3. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <200 c/mL at Week 96
Description: Percentage of participants with plasma HIV-1 RNA <200 c/mL was assessed at Week 96 according to the FDA snapshot algorithm.
Time Frame: Week 96
Population: Intent To Treat-Exposed
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Percentage of Participants | 69 [50 to 84]

4. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <200 c/mL at Week 144
Description: Percentage of participants with plasma HIV-1 RNA <200 c/mL was assessed at Week 144 according to the FDA snapshot algorithm.
Time Frame: Week 144
Population: Intent To Treat-Exposed
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Percentage of Participants | 66 [47 to 81]

5. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Week 24
Description: Percentage of participants with plasma HIV-1 RNA <50 c/mL was assessed at Week 24 according to the FDA snapshot algorithm.
Time Frame: Week 24
Population: Intent To Treat-Exposed
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Percentage of Participants | 84 [67 to 95]

6. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Week 96
Description: Percentage of participants with plasma HIV-1 RNA <50 c/mL was assessed at Week 96 according to the FDA snapshot algorithm.
Time Frame: Week 96
Population: Intent To Treat-Exposed
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Percentage of Participants | 69 [50 to 84]

7. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Week 144
Description: Percentage of participants with plasma HIV-1 RNA <50 c/mL was assessed at Week 144 according to the FDA Snapshot algorithm.
Time Frame: Week 144
Population: Intent To Treat-Exposed
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Percentage of Participants | 66 [47 to 81]

8. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <200 c/mL at Week 48
Description: Percentage of participants with plasma HIV-1 RNA <200 c/mL was assessed at Week 48 according to the FDA snapshot algorithm.
Time Frame: Week 48
Population: Intent To Treat-Exposed
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Percentage of Participants | 84 [67 to 95]

9. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) Through 144 Weeks
Description: An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A serious adverse event is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment.
Time Frame: Up to 144 weeks
Population: Safety population includes participants who have received at least one dose of DTG/3TC.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  AEs | 29
  SAEs | 5

10. Secondary Outcome: Number of Participants With AEs Through 144 Weeks by Severity
Description: The Division of Acquired Immunodeficiency Syndrome (DAIDS) criteria for grading the severity of adult and pediatric adverse events was used to assess severity. Grades were defined based on numeric criteria as follows: Grade 1 - mild; Grade 2 - moderate; Grade 3 - severe or medically significant; Grade 4 - life-threatening consequences; Grade 5 - death. A higher grade indicates a greater severity.
Time Frame: Up to 144 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  Grade 1 | 5
  Grade 2 | 19
  Grade 3 | 5
  Grade 4 | 0
  Grade 5 | 0

11. Secondary Outcome: Number of Participants With Abnormal Findings for Hematology Parameters Through 144 Weeks
Description: Blood samples were collected from participants for analysis of hematology parameters including hemoglobin, leukocytes and neutrophils. The DAIDS criteria for grading the severity of adult and pediatric adverse events was used to assess severity. Grades were defined based on numeric criteria as follows: Grade 0 - no abnormality; Grade 1 - mild; Grade 2 - moderate; Grade 3 - severe or medically significant; Grade 4 - life-threatening consequences.
Time Frame: Up to 144 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  Hemoglobin: Grade 1 | 0
  Hemoglobin: Grade 2 | 4
  Hemoglobin: Grade 3 | 0
  Hemoglobin: Grade 4 | 0
  Hemoglobin: Grade 0 | 28
  Leukocytes: Grade 1 | 2
  Leukocytes: Grade 2 | 0
  Leukocytes: Grade 3 | 0
  Leukocytes: Grade 4 | 0
  Leukocytes: Grade 0 | 30
  Neutrophils: Grade 1 | 0
  Neutrophils: Grade 2 | 1
  Neutrophils: Grade 3 | 0
  Neutrophils: Grade 4 | 0
  Neutrophils: Grade 0 | 31

12. Secondary Outcome: Number of Participants With Abnormal Findings for Clinical Chemistry Parameters Through 144 Weeks
Description: Blood samples were collected from participants for analysis of clinical chemistry parameters including potassium, aspartate aminotransferase, creatinine, alanine aminotransferase (ALT), carbon dioxide, alkaline phosphatase, bilirubin, direct bilirubin, sodium, GFR from creatinine adjusted for BSA, calcium, and creatine kinase. Grades were defined based on numeric criteria as follows: Grade 0 - no abnormality; Grade 1 - mild; Grade 2 - moderate; Grade 3 - severe or medically significant; Grade 4 - life-threatening consequences.
Time Frame: Up to 144 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  Alanine Aminotransferase: Grade 1 | 3
  Alanine Aminotransferase: Grade 2 | 1
  Alanine Aminotransferase: Grade 3 | 0
  Alanine Aminotransferase: Grade 4 | 0
  Alanine Aminotransferase: Grade 0 | 28
  Alkaline Phosphatase: Grade 1 | 1
  Alkaline Phosphatase: Grade 2 | 2
  Alkaline Phosphatase: Grade 3 | 0
  Alkaline Phosphatase: Grade 4 | 0
  Alkaline Phosphatase: Grade 0 | 29
  Aspartate Aminotransferase: Grade 1 | 2
  Aspartate Aminotransferase: Grade 2 | 0
  Aspartate Aminotransferase: Grade 3 | 0
  Aspartate Aminotransferase: Grade 4 | 0
  Aspartate Aminotransferase: Grade 0 | 30
  Bilirubin: Grade 1 | 1
  Bilirubin: Grade 2 | 1
  Bilirubin: Grade 3 | 0
  Bilirubin: Grade 4 | 0
  Bilirubin: Grade 0 | 30
  Calcium: Grade 1 | 0
  Calcium: Grade 2 | 1
  Calcium: Grade 3 | 0
  Calcium: Grade 4 | 1
  Calcium: Grade 0 | 30
  Carbon Dioxide: Grade 1 | 17
  Carbon Dioxide: Grade 2 | 5
  Carbon Dioxide: Grade 3 | 0
  Carbon Dioxide: Grade 4 | 2
  Carbon Dioxide: Grade 0 | 8
  Creatine Kinase: Grade 1 | 2
  Creatine Kinase: Grade 2 | 2
  Creatine Kinase: Grade 3 | 2
  Creatine Kinase: Grade 4 | 0
  Creatine Kinase: Grade 0 | 26
  Creatinine: Grade 1 | 2
  Creatinine: Grade 2 | 0
  Creatinine: Grade 3 | 0
  Creatinine: Grade 4 | 0
  Creatinine: Grade 0 | 30
  Direct Bilirubin: Grade 1 | 0
  Direct Bilirubin: Grade 2 | 0
  Direct Bilirubin: Grade 3 | 1
  Direct Bilirubin: Grade 4 | 0
  Direct Bilirubin: Grade 0 | 31
  GFR from Creatinine Adjusted for BSA: Grade 1 | 0
  GFR from Creatinine Adjusted for BSA: Grade 2 | 14
  GFR from Creatinine Adjusted for BSA: Grade 3 | 5
  GFR from Creatinine Adjusted for BSA: Grade 4 | 0
  GFR from Creatinine Adjusted for BSA: Grade 0 | 13
  Potassium: Grade 1 | 2
  Potassium: Grade 2 | 0
  Potassium: Grade 3 | 0
  Potassium: Grade 4 | 0
  Potassium: Grade 0 | 30
  Sodium: Grade 1 | 6
  Sodium: Grade 2 | 1
  Sodium: Grade 3 | 0
  Sodium: Grade 4 | 0
  Sodium: Grade 0 | 25

13. Secondary Outcome: Number of Participants With Abnormal Findings for Fasting Lipids Through 144 Weeks
Description: Lipid assessments including cholesterol, low density lipoprotein (LDL) cholesterol, LDL Cholesterol Calculation, LDL Cholesterol Direct, and triglycerides were performed. Grades were defined based on numeric criteria as follows: Grade 0 - no abnormality; Grade 1 - mild; Grade 2 - moderate; Grade 3 - severe or medically significant; Grade 4 - life-threatening consequences.
Time Frame: Up to 144 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  Cholesterol: Grade 1 | 7
  Cholesterol: Grade 2 | 1
  Cholesterol: Grade 3 | 0
  Cholesterol: Grade 4 | 0
  Cholesterol: Grade 0 | 24
  LDL Cholesterol: Grade 1 | 2
  LDL Cholesterol: Grade 2 | 0
  LDL Cholesterol: Grade 3 | 0
  LDL Cholesterol: Grade 4 | 0
  LDL Cholesterol: Grade 0 | 30
  LDL Cholesterol Calculation: Grade 1 | 2
  LDL Cholesterol Calculation: Grade 2 | 0
  LDL Cholesterol Calculation: Grade 3 | 0
  LDL Cholesterol Calculation: Grade 4 | 0
  LDL Cholesterol Calculation: Grade 0 | 30
  LDL Cholesterol Direct: Grade 1 | 6
  LDL Cholesterol Direct: Grade 2 | 3
  LDL Cholesterol Direct: Grade 3 | 0
  LDL Cholesterol Direct: Grade 4 | 0
  LDL Cholesterol Direct: Grade 0 | 23
  Triglycerides: Grade 1 | 5
  Triglycerides: Grade 2 | 0
  Triglycerides: Grade 3 | 0
  Triglycerides: Grade 4 | 0
  Triglycerides: Grade 0 | 27

14. Secondary Outcome: Number of Participants With Abnormal Findings for Urinalysis Parameters Through 144 Weeks
Description: Urine samples were collected from participants for the analysis of urinalysis parameters including urinary glucose, urinary protein, and urine erythrocytes. Grades were defined based on numeric criteria as follows: Grade 0 - no abnormality; Grade 1 - mild; Grade 2 - moderate; Grade 3 - severe or medically significant; Grade 4 - life-threatening consequences.
Time Frame: Up to 144 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  Urinary Glucose: Grade 1 | 1
  Urinary Glucose: Grade 2 | 0
  Urinary Glucose: Grade 3 | 0
  Urinary Glucose: Grade 4 | 0
  Urinary Glucose: Grade 0 | 31
  Urinary Protein: Grade 1 | 5
  Urinary Protein: Grade 2 | 2
  Urinary Protein: Grade 3 | 0
  Urinary Protein: Grade 4 | 0
  Urinary Protein: Grade 0 | 25
  Urine Erythrocytes: Grade 1 | 2
  Urine Erythrocytes: Grade 2 | 0
  Urine Erythrocytes: Grade 3 | 0
  Urine Erythrocytes: Grade 4 | 0
  Urine Erythrocytes: Grade 0 | 30

15. Secondary Outcome: Number of Participants Who Discontinue Treatment Due to Adverse Events Through 144 Weeks
Time Frame: Up to 144 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants | 2

16. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events Through 96 Weeks
Time Frame: Up to 96 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  AEs | 29
  SAEs | 3

17. Secondary Outcome: Number of Participants With Severity of Adverse Events Through 96 Weeks
Description: AEs were evaluated by the investigator and graded according to the DAIDS toxicity scales as follows: Grade 1 - mild; Grade 2 - moderate; Grade 3 - severe or medically significant; Grade 4 - life-threatening consequences; Grade 5 - death. The higher the grade, the more severe the symptoms.
Time Frame: Up to 96 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  Grade 1 | 8
  Grade 2 | 19
  Grade 3 | 2
  Grade 4 | 0
  Grade 5 | 0

18. Secondary Outcome: Number of Participants With Abnormal Findings for Hematology Parameters Through 96 Weeks
Description: Blood samples were collected from participants for analysis of hematology parameters including hemoglobin, leukocytes and neutrophils. Grades were defined based on numeric criteria as follows: Grade 0 - no abnormality; Grade 1 - mild; Grade 2 - moderate; Grade 3 - severe or medically significant; Grade 4 - life-threatening consequences.
Time Frame: Up to 96 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  Hemoglobin: Grade 1 | 0
  Hemoglobin: Grade 2 | 4
  Hemoglobin: Grade 3 | 0
  Hemoglobin: Grade 4 | 0
  Hemoglobin: Grade 0 | 28
  Leukocytes: Grade 1 | 2
  Leukocytes: Grade 2 | 0
  Leukocytes: Grade 3 | 0
  Leukocytes: Grade 4 | 0
  Leukocytes: Grade 0 | 30
  Neutrophils: Grade 1 | 0
  Neutrophils: Grade 2 | 1
  Neutrophils: Grade 3 | 0
  Neutrophils: Grade 4 | 0
  Neutrophils: Grade 0 | 31

19. Secondary Outcome: Number of Participants With Abnormal Findings for Clinical Chemistry Parameters Through 96 Weeks
Description: Blood samples were collected from participants for analysis of clinical chemistry parameters including potassium, aspartate aminotransferase, creatinine, alanine aminotransferase, carbon dioxide, alkaline phosphatase, bilirubin, sodium, GFR from creatinine adjusted for BSA, calcium, and creatine kinase. Grades were defined based on numeric criteria as follows: Grade 0 - no abnormality; Grade 1 - mild; Grade 2 - moderate; Grade 3 - severe or medically significant; Grade 4 - life-threatening consequences.
Time Frame: Up to 96 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  Alanine Aminotransferase: Grade 1 | 2
  Alanine Aminotransferase: Grade 2 | 1
  Alanine Aminotransferase: Grade 3 | 0
  Alanine Aminotransferase: Grade 4 | 0
  Alanine Aminotransferase: Grade 0 | 29
  Alkaline Phosphatase: Grade 1 | 1
  Alkaline Phosphatase: Grade 2 | 2
  Alkaline Phosphatase: Grade 3 | 0
  Alkaline Phosphatase: Grade 4 | 0
  Alkaline Phosphatase: Grade 0 | 29
  Aspartate Aminotransferase: Grade 1 | 2
  Aspartate Aminotransferase: Grade 2 | 0
  Aspartate Aminotransferase: Grade 3 | 0
  Aspartate Aminotransferase: Grade 4 | 0
  Aspartate Aminotransferase: Grade 0 | 30
  Bilirubin: Grade 1 | 2
  Bilirubin: Grade 2 | 0
  Bilirubin: Grade 3 | 0
  Bilirubin: Grade 4 | 0
  Bilirubin: Grade 0 | 30
  Calcium: Grade 1 | 0
  Calcium: Grade 2 | 1
  Calcium: Grade 3 | 0
  Calcium: Grade 4 | 1
  Calcium: Grade 0 | 30
  Carbon Dioxide: Grade 1 | 14
  Carbon Dioxide: Grade 2 | 5
  Carbon Dioxide: Grade 3 | 0
  Carbon Dioxide: Grade 4 | 2
  Carbon Dioxide: Grade 0 | 11
  Creatine Kinase: Grade 1 | 2
  Creatine Kinase: Grade 2 | 1
  Creatine Kinase: Grade 3 | 2
  Creatine Kinase: Grade 4 | 0
  Creatine Kinase: Grade 0 | 27
  Creatinine: Grade 1 | 2
  Creatinine: Grade 2 | 0
  Creatinine: Grade 3 | 0
  Creatinine: Grade 4 | 0
  Creatinine: Grade 0 | 30
  GFR from Creatinine Adjusted for BSA: Grade 1 | 0
  GFR from Creatinine Adjusted for BSA: Grade 2 | 13
  GFR from Creatinine Adjusted for BSA: Grade 3 | 5
  GFR from Creatinine Adjusted for BSA: Grade 4 | 0
  GFR from Creatinine Adjusted for BSA: Grade 0 | 14
  Potassium: Grade 1 | 2
  Potassium: Grade 2 | 0
  Potassium: Grade 3 | 0
  Potassium: Grade 4 | 0
  Potassium: Grade 0 | 30
  Sodium: Grade 1 | 5
  Sodium: Grade 2 | 1
  Sodium: Grade 3 | 0
  Sodium: Grade 4 | 0
  Sodium: Grade 0 | 26

20. Secondary Outcome: Number of Participants With Abnormal Findings for Fasting Lipids Through 96 Weeks
Description: Lipid assessments including cholesterol, LDL cholesterol, LDL cholesterol calculation, LDL cholesterol direct, and triglycerides were performed. Grades were defined based on numeric criteria as follows: Grade 0 - no abnormality; Grade 1 - mild; Grade 2 - moderate; Grade 3 - severe or medically significant; Grade 4 - life-threatening consequences.
Time Frame: Up to 96 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  Cholesterol: Grade 1 | 7
  Cholesterol: Grade 2 | 1
  Cholesterol: Grade 3 | 0
  Cholesterol: Grade 4 | 0
  Cholesterol: Grade 0 | 24
  LDL Cholesterol: Grade 1 | 2
  LDL Cholesterol: Grade 2 | 0
  LDL Cholesterol: Grade 3 | 0
  LDL Cholesterol: Grade 4 | 0
  LDL Cholesterol: Grade 0 | 30
  LDL Cholesterol Calculation: Grade 1 | 1
  LDL Cholesterol Calculation: Grade 2 | 0
  LDL Cholesterol Calculation: Grade 3 | 0
  LDL Cholesterol Calculation: Grade 4 | 0
  LDL Cholesterol Calculation: Grade 0 | 31
  LDL Cholesterol Direct: Grade 1 | 6
  LDL Cholesterol Direct: Grade 2 | 2
  LDL Cholesterol Direct: Grade 3 | 0
  LDL Cholesterol Direct: Grade 4 | 0
  LDL Cholesterol Direct: Grade 0 | 24
  Triglycerides: Grade 1 | 4
  Triglycerides: Grade 2 | 0
  Triglycerides: Grade 3 | 0
  Triglycerides: Grade 4 | 0
  Triglycerides: Grade 0 | 28

21. Secondary Outcome: Number of Participants With Abnormal Findings for Urinalysis Parameters Through 96 Weeks
Description: Urine samples will be collected from participants for the analysis of urinalysis parameters including urinary glucose, urinary protein, and urine erythrocytes. Grades were defined based on numeric criteria as follows: Grade 0 - no abnormality; Grade 1 - mild; Grade 2 - moderate; Grade 3 - severe or medically significant; Grade 4 - life-threatening consequences.
Time Frame: Up to 96 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  Urinary Glucose: Grade 1 | 1
  Urinary Glucose: Grade 2 | 0
  Urinary Glucose: Grade 3 | 0
  Urinary Glucose: Grade 4 | 0
  Urinary Glucose: Grade 0 | 31
  Urinary Protein: Grade 1 | 3
  Urinary Protein: Grade 2 | 2
  Urinary Protein: Grade 3 | 0
  Urinary Protein: Grade 4 | 0
  Urinary Protein: Grade 0 | 27
  Urine Erythrocytes: Grade 1 | 2
  Urine Erythrocytes: Grade 2 | 0
  Urine Erythrocytes: Grade 3 | 0
  Urine Erythrocytes: Grade 4 | 0
  Urine Erythrocytes: Grade 0 | 30

22. Secondary Outcome: Number of Participants Undergoing Viral Load Monitoring From Week 48 Through 144 Weeks
Description: Viral load was defined as plasma HIV-RNA <50 copies per mL. Viral load monitoring of participants was performed from Week 48 through 144 weeks.
Time Frame: Weeks 48, 60, 72, 84, 96, 108, 120, 132, and 144
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  Week 48 | 28
  Week 60 | 27
  Week 72 | 23
  Week 84 | 23
  Week 96 | 23
  Week 108 | 21
  Week 120 | 21
  Week 132 | 21
  Week 144 | 21

23. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4+ (CD4+) Cell Count at Weeks 24 and 48
Description: Baseline value was defined as the latest pre-dose assessment with a non-missing value (Day 1). Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 24 and 48
Population: Intent-To-Treat Exposed. Only those participants with data available at specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: 10^6 cells per liter
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
10^6 cells per liter
  Baseline (Day 1) | 371.500 [270.00 to 507.50]
  Week 24: number analyzed (Participants) | 29
  Week 24 | 167.000 [103.00 to 319.00]
  Week 48: number analyzed (Participants) | 28
  Week 48 | 223.500 [85.50 to 380.50]

24. Secondary Outcome: Change From Baseline in CD8+ Cell Count at Weeks 24 and 48
Description: as for outcome 23
Time Frame: Baseline (Day 1) and Weeks 24 and 48
Population: Intent-To-Treat Exposed. Only those participants with data available at specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: 10^6 cells per liter
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
10^6 cells per liter
  Baseline (Day 1) | 828.000 [679.50 to 1031.50]
  Week 24: number analyzed (Participants) | 29
  Week 24 | -15.000 [-117.00 to 301.00]
  Week 48: number analyzed (Participants) | 28
  Week 48 | -78.500 [-243.00 to 176.00]

25. Secondary Outcome: Change From Baseline in Ratio of CD4+ and CD8+ at Weeks 24 and 48
Description: as for outcome 23
Time Frame: Baseline (Day 1) and Weeks 24 and 48
Population: Intent-To-Treat Exposed. Only those participants with data available at specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Ratio
  Baseline (Day 1) | 0.395 [0.33 to 0.64]
  Week 24: number analyzed (Participants) | 26
  Week 24 | 0.215 [0.14 to 0.30]
  Week 48: number analyzed (Participants) | 28
  Week 48 | 0.345 [0.24 to 0.49]

26. Secondary Outcome: Number of Participants With Disease Progression From Week 24 Through Week 48
Description: Participants with disease progression included incidences of HIV-associated conditions, Acquired Immuno Deficiency Syndrome (AIDS) and death. HIV-associated conditions were assessed according to the 2014 HIV infection by Centers for Disease Control and Prevention (CDC) classification system for HIV Infection in adults to evaluate the immune effects of DTG /3TC FDC.
Time Frame: Week 24 and up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  Week 24 | 0
  Week 48 | 1

27. Secondary Outcome: Number of Participants With Any Adverse Events and Serious Adverse Events From Week 24 Through Week 48
Time Frame: Week 24 and up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  AEs (Week 24) | 23
  AEs (Week 48) | 28
  SAEs (Week 24) | 1
  SAEs (Week 48) | 2

28. Secondary Outcome: Number of Participants With Severity of Adverse Events From Week 24 Through Week 48
Description: as for outcome 17
Time Frame: Week 24 and up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  Grade 1 (Week 24) | 9
  Grade 2 (Week 24) | 13
  Grade 3 (Week 24) | 1
  Grade 4 (Week 24) | 0
  Grade 5 (Week 24) | 0
  Grade 1 (Week 48) | 11
  Grade 2 (Week 48) | 16
  Grade 3 (Week 48) | 1
  Grade 4 (Week 48) | 0
  Grade 5 (Week 48) | 0

29. Secondary Outcome: Number of Participants With Abnormal Findings for Hematology Parameters From Week 24 Through Week 48
Description: Blood samples were collected from participants for analysis of hematology parameters including hemoglobin, leukocytes and neutrophils. Grades were defined based on numeric criteria as follows: Grade 1 - mild; Grade 2 - moderate; Grade 3 - severe or medically significant; Grade 4 - life-threatening consequences.
Time Frame: Week 24 and up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  Hemoglobin - Grade 1 (Week 24) | 0
  Hemoglobin - Grade 2 (Week 24) | 2
  Hemoglobin - Grade 3 (Week 24) | 0
  Hemoglobin - Grade 4 (Week 24) | 0
  Leukocytes - Grade 1 (Week 24) | 1
  Leukocytes - Grade 2 (Week 24) | 0
  Leukocytes - Grade 3 (Week 24) | 0
  Leukocytes - Grade 4 (Week 24) | 0
  Neutrophils - Grade 1 (Week 24) | 0
  Neutrophils - Grade 2 (Week 24) | 1
  Neutrophils - Grade 3 (Week 24) | 0
  Neutrophils - Grade 4 (Week 24) | 0
  Hemoglobin - Grade 1 (Week 48) | 0
  Hemoglobin - Grade 2 (Week 48) | 2
  Hemoglobin - Grade 3 (Week 48) | 0
  Hemoglobin - Grade 4 (Week 48) | 0
  Leukocytes - Grade 1 (Week 48) | 2
  Leukocytes - Grade 2 (Week 48) | 0
  Leukocytes - Grade 3 (Week 48) | 0
  Leukocytes - Grade 4 (Week 48) | 0
  Neutrophils - Grade 1 (Week 48) | 0
  Neutrophils - Grade 2 (Week 48) | 1
  Neutrophils - Grade 3 (Week 48) | 0
  Neutrophils - Grade 4 (Week 48) | 0

30. Secondary Outcome: Number of Participants With Abnormal Findings for Clinical Chemistry Parameters From Week 24 Through Week 48
Description: Blood samples were collected from participants for analysis of clinical chemistry parameters including potassium, aspartate aminotransferase, creatinine, alanine aminotransferase, carbon dioxide, alkaline phosphatase, bilirubin, sodium, GFR from creatinine adjusted for BSA, calcium, and creatine kinase. Grades were defined based on numeric criteria as follows: Grade 1 - mild; Grade 2 - moderate; Grade 3 - severe or medically significant; Grade 4 - life-threatening consequences.
Time Frame: Week 24 and up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  Alanine Aminotransferase - Grade 1 (Week 24) | 1
  Alanine Aminotransferase - Grade 2 (Week 24) | 0
  Alanine Aminotransferase - Grade 3 (Week 24) | 0
  Alanine Aminotransferase - Grade 4 (Week 24) | 0
  Alkaline Phosphatase - Grade 1 (Week 24) | 1
  Alkaline Phosphatase - Grade 2 (Week 24) | 2
  Alkaline Phosphatase - Grade 3 (Week 24) | 0
  Alkaline Phosphatase - Grade 4 (Week 24) | 0
  Aspartate Aminotransferase - Grade 1 (Week 24) | 1
  Aspartate Aminotransferase - Grade 2 (Week 24) | 0
  Aspartate Aminotransferase - Grade 3 (Week 24) | 0
  Aspartate Aminotransferase - Grade 4 (Week 24) | 0
  Bilirubin - Grade 1 (Week 24) | 1
  Bilirubin - Grade 2 (Week 24) | 0
  Bilirubin - Grade 3 (Week 24) | 0
  Bilirubin - Grade 4 (Week 24) | 0
  Calcium - Grade 1 (Week 24) | 0
  Calcium - Grade 2 (Week 24) | 1
  Calcium - Grade 3 (Week 24) | 0
  Calcium - Grade 4 (Week 24) | 1
  Carbon Dioxide - Grade 1 (Week 24) | 11
  Carbon Dioxide - Grade 2 (Week 24) | 4
  Carbon Dioxide - Grade 3 (Week 24) | 0
  Carbon Dioxide - Grade 4 (Week 24) | 2
  Creatine Kinase - Grade 1 (Week 24) | 1
  Creatine Kinase - Grade 2 (Week 24) | 0
  Creatine Kinase - Grade 3 (Week 24) | 0
  Creatine Kinase - Grade 4 (Week 24) | 0
  Creatinine - Grade 1 (Week 24) | 1
  Creatinine - Grade 2 (Week 24) | 0
  Creatinine - Grade 3 (Week 24) | 0
  Creatinine - Grade 4 (Week 24) | 0
  GFR from Creatinine Adjusted for BSA - Grade 1 (Week 24) | 0
  GFR from Creatinine Adjusted for BSA - Grade 2 (Week 24) | 12
  GFR from Creatinine Adjusted for BSA - Grade 3 (Week 24) | 3
  GFR from Creatinine Adjusted for BSA - Grade 4 (Week 24) | 0
  Potassium - Grade 1 (Week 24) | 1
  Potassium - Grade 2 (Week 24) | 0
  Potassium - Grade 3 (Week 24) | 0
  Potassium - Grade 4 (Week 24) | 0
  Sodium - Grade 1 (Week 24) | 5
  Sodium - Grade 2 (Week 24) | 1
  Sodium - Grade 3 (Week 24) | 0
  Sodium - Grade 4 (Week 24) | 0
  Alanine Aminotransferase - Grade 1 (Week 48) | 1
  Alanine Aminotransferase - Grade 2 (Week 48) | 0
  Alanine Aminotransferase - Grade 3 (Week 48) | 0
  Alanine Aminotransferase - Grade 4 (Week 48) | 0
  Alkaline Phosphatase - Grade 1 (Week 48) | 1
  Alkaline Phosphatase - Grade 2 (Week 48) | 2
  Alkaline Phosphatase - Grade 3 (Week 48) | 0
  Alkaline Phosphatase - Grade 4 (Week 48) | 0
  Aspartate Aminotransferase - Grade 1 (Week 48) | 1
  Aspartate Aminotransferase - Grade 2 (Week 48) | 0
  Aspartate Aminotransferase - Grade 3 (Week 48) | 0
  Aspartate Aminotransferase - Grade 4 (Week 48) | 0
  Bilirubin - Grade 1 (Week 48) | 1
  Bilirubin - Grade 2 (Week 48) | 0
  Bilirubin - Grade 3 (Week 48) | 0
  Bilirubin - Grade 4 (Week 48) | 0
  Calcium - Grade 1 (Week 48) | 0
  Calcium - Grade 2 (Week 48) | 1
  Calcium - Grade 3 (Week 48) | 0
  Calcium - Grade 4 (Week 48) | 1
  Carbon Dioxide - Grade 1 (Week 48) | 12
  Carbon Dioxide - Grade 2 (Week 48) | 5
  Carbon Dioxide - Grade 3 (Week 48) | 0
  Carbon Dioxide - Grade 4 (Week 48) | 2
  Creatine Kinase - Grade 1 (Week 48) | 1
  Creatine Kinase - Grade 2 (Week 48) | 0
  Creatine Kinase - Grade 3 (Week 48) | 0
  Creatine Kinase - Grade 4 (Week 48) | 0
  Creatinine - Grade 1 (Week 48) | 2
  Creatinine - Grade 2 (Week 48) | 0
  Creatinine - Grade 3 (Week 48) | 0
  Creatinine - Grade 4 (Week 48) | 0
  GFR from Creatinine Adjusted for BSA - Grade 1 (Week 48) | 0
  GFR from Creatinine Adjusted for BSA - Grade 2 (Week 48) | 13
  GFR from Creatinine Adjusted for BSA - Grade 3 (Week 48) | 6
  GFR from Creatinine Adjusted for BSA - Grade 4 (Week 48) | 0
  Potassium - Grade 1 (Week 48) | 1
  Potassium - Grade 2 (Week 48) | 0
  Potassium - Grade 3 (Week 48) | 0
  Potassium - Grade 4 (Week 48) | 0
  Sodium - Grade 1 (Week 48) | 5
  Sodium - Grade 2 (Week 48) | 1
  Sodium - Grade 3 (Week 48) | 0
  Sodium - Grade 4 (Week 48) | 0

31. Secondary Outcome: Number of Participants With Abnormal Findings for Fasting Lipids From Week 24 Through Week 48
Description: Lipid assessments including cholesterol, LDL cholesterol, LDL cholesterol calculation, LDL cholesterol direct, and triglycerides were performed. Grades were defined based on numeric criteria as follows: Grade 1 - mild; Grade 2 - moderate; Grade 3 - severe or medically significant; Grade 4 - life-threatening consequences.
Time Frame: Week 24 and up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  Cholesterol - Grade 1 (Week 24) | 2
  Cholesterol - Grade 2 (Week 24) | 0
  Cholesterol - Grade 3 (Week 24) | 0
  Cholesterol - Grade 4 (Week 24) | 0
  LDL cholesterol - Grade 1 (Week 24) | 1
  LDL cholesterol - Grade 2 (Week 24) | 0
  LDL cholesterol - Grade 3 (Week 24) | 0
  LDL cholesterol - Grade 4 (Week 24) | 0
  Triglycerides - Grade 1 (Week 24) | 1
  Triglycerides - Grade 2 (Week 24) | 0
  Triglycerides - Grade 3 (Week 24) | 0
  Triglycerides - Grade 4 (Week 24) | 0
  Cholesterol - Grade 1 (Week 48) | 5
  Cholesterol - Grade 2 (Week 48) | 1
  Cholesterol - Grade 3 (Week 48) | 0
  Cholesterol - Grade 4 (Week 48) | 0
  LDL cholesterol - Grade 1 (Week 48) | 1
  LDL cholesterol - Grade 2 (Week 48) | 0
  LDL cholesterol - Grade 3 (Week 48) | 0
  LDL cholesterol - Grade 4 (Week 48) | 0
  Triglycerides - Grade 1 (Week 48) | 1
  Triglycerides - Grade 2 (Week 48) | 0
  Triglycerides - Grade 3 (Week 48) | 0
  Triglycerides - Grade 4 (Week 48) | 0

32. Secondary Outcome: Number of Participants With Abnormal Findings for Urinalysis Parameters From Week 24 Through Week 48
Description: Urine samples will be collected from participants for the analysis of urinalysis parameters including urinary glucose, urinary protein, and urine erythrocytes. Grades were defined based on numeric criteria as follows: Grade 1 - mild; Grade 2 - moderate; Grade 3 - severe or medically significant; Grade 4 - life-threatening consequences.
Time Frame: Week 24 and up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  Urinary Glucose - Grade 1 (Week 24) | 0
  Urinary Glucose - Grade 2 (Week 24) | 0
  Urinary Glucose - Grade 3 (Week 24) | 0
  Urinary Glucose - Grade 4 (Week 24) | 0
  Urinary Protein - Grade 1 (Week 24) | 0
  Urinary Protein - Grade 2 (Week 24) | 0
  Urinary Protein - Grade 3 (Week 24) | 0
  Urinary Protein - Grade 4 (Week 24) | 0
  Urinary Glucose - Grade 1 (Week 48) | 1
  Urinary Glucose - Grade 2 (Week 48) | 0
  Urinary Glucose - Grade 3 (Week 48) | 0
  Urinary Glucose - Grade 4 (Week 48) | 0
  Urinary Protein - Grade 1 (Week 48) | 1
  Urinary Protein - Grade 2 (Week 48) | 1
  Urinary Protein - Grade 3 (Week 48) | 0
  Urinary Protein - Grade 4 (Week 48) | 0

33. Secondary Outcome: Number of Participants Who Discontinued Treatment Due to Adverse Events From Week 24 Through Week 48
Time Frame: Week 24 and up to Week 48
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 32
Participants
  Week 24 | 1
  Week 48 | 1

34. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Dosing With DTG and 3TC
Description: Blood samples were collected on a subset of participants for intensive pharmacokinetic analysis.
Time Frame: Pre-dose, 0.5, 1.0, 1.5, 2, 3, 4, 6, 10, and 24 hours post-dose at Week 1
Population: Intensive Pharmacokinetic Population includes all participants who received at least 1 dose of DTG/3TC FDC and have evaluable drug concentrations reported, where samples are collected according to the intensive sampling schedule.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 12
Nanogram per milliliter (ng/mL)
  Maximum observed plasma concentration - DTG | 5354.870 (25.02)
  Maximum observed plasma concentration - 3TC | 2778.555 (27.80)

35. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) Following Dosing With DTG and 3TC
Description: Blood samples were collected on a subset of participants for intensive pharmacokinetic analysis.
Time Frame: Pre-dose, 0.5, 1.0, 1.5, 2, 3, 4, 6, 10, and 24 hours post-dose at Week 1
Population: Intensive Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 12
Hours
  Time of maximum observed plasma concentration - DTG | 2.000 [1.00 to 3.00]
  Time of maximum observed plasma concentration - 3TC | 1.000 [1.00 to 3.00]

36. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration (AUC[0-t]) Following Dosing With DTG and 3TC
Description: Blood samples were collected on a subset of participants for intensive pharmacokinetic analysis.
Time Frame: Pre-dose, 0.5, 1.0, 1.5, 2, 3, 4, 6, 10, and 24 hours post-dose at Week 1
Population: Intensive Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 12
hours*nanogram per milliliter (h*ng/mL)
  AUC[0-t] - DTG | 74001.76 (23.2)
  AUC[0-t] - 3TC | 12277.62 (17.7)

37. Secondary Outcome: Area Under the Curve (AUC) Over the Dosing Interval (AUC[0-tau]) Following Dosing With DTG and 3TC
Description: Blood samples were collected on a subset of participants for intensive pharmacokinetic analysis.
Time Frame: Pre-dose, 0.5, 1.0, 1.5, 2, 3, 4, 6, 10, and 24 hours post-dose at Week 1
Population: Intensive Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 12
hours*nanogram per milliliter (h*ng/mL)
  AUC[0-tau] - DTG | 74001.76 (23.2)
  AUC[0-tau] - 3TC | 12277.62 (17.7)

38. Secondary Outcome: Apparent Terminal Half-life (t1/2) Following Dosing With DTG and 3TC
Description: Blood samples were collected on a subset of participants for intensive pharmacokinetic analysis.
Time Frame: Pre-dose, 0.5, 1.0, 1.5, 2, 3, 4, 6, 10, and 24 hours post-dose at Week 1
Population: Intensive Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 12
Hours
  Apparent terminal half-life - DTG | 12.910 (15.35)
  Apparent terminal half-life - 3TC | 4.823 (13.26)

39. Secondary Outcome: Observed Pre-dose Plasma Concentration Following Dosing With DTG and 3TC
Description: Blood samples were collected on a subset of participants for intensive pharmacokinetic analysis.
Time Frame: Pre-dose at Week 1
Population: Intensive Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 12
ng/mL
  DTG | 1636.791 (39.26)
  3TC | 51.073 (60.88)

40. Secondary Outcome: Observed Plasma Concentration at 24 Hours Following Dosing With DTG and 3TC
Description: Blood samples were collected on a subset of participants for intensive pharmacokinetic analysis.
Time Frame: 24 hours post-dose at Week 1
Population: Intensive Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 12
ng/mL
  DTG | 1635.606 (25.36)
  3TC | 53.453 (33.42)

41. Secondary Outcome: Number of Participants With Observed Genotypic Resistance to DTG and 3TC
Description: Protocol-defined confirmed virologic withdrawal (CVW) through Week 144 was low with 1 participant meeting CVW criteria. Resistance testing failed, and therefore no genotypic data were available for this participant at the time of virologic failure.
Time Frame: Up to 144 weeks
Population: The analysis used the CVW population, comprising ITT-E participants meeting CVW criteria: confirmed virologic non-response (HIV-1 RNA <1 log10 c/mL at/after Week 12 or =200 c/mL at/after Week 24) or confirmed rebound (HIV-1 RNA =200 c/mL after prior suppression <200 c/mL).
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 1
Participants | 0

42. Secondary Outcome: Number of Participants With Observed Phenotypic Resistance to DTG and 3TC
Description: Protocol-defined CVW through Week 144 was low with 1 participant meeting CVW criteria. Resistance testing failed, and therefore no phenotypic data were available for this participant at the time of virologic failure.
Time Frame: Up to 144 weeks
Population: CVW Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG/3TC FDC
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: All-Cause mortality, Non-SAEs and SAEs were collected from Day 1 up to Week 144
Arm/Group | DTG/3TC FDC
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 5/32
Other Adverse Events (participants affected / at risk) | 29/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG/3TC FDC (N=32)
Anal abscess (Infections and infestations) | 1 (1)
Vulvovaginal warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Orchitis (Infections and infestations) | 1 (1)
Ulcerative keratitis (Eye disorders) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG/3TC FDC (N=32)
Nasopharyngitis (Infections and infestations) | 8 (10)
Folliculitis (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 6 (7)
Genital herpes (Infections and infestations) | 2 (2)
Pharyngitis (Infections and infestations) | 5 (5)
Vulvovaginal candidiasis (Infections and infestations) | 2 (2)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (5)
COVID-19 (Infections and infestations) | 10 (16)
Herpes zoster (Infections and infestations) | 2 (2)
Tonsillitis (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2)
Aphthous ulcer (Gastrointestinal disorders) | 2 (3)
Food poisoning (Gastrointestinal disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypersensitivity (Immune system disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Depression (Psychiatric disorders) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2)
Glomerular filtration rate decreased (Investigations) | 2 (3)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Secondary syphilis (Infections and infestations) | 3 (4)
Impetigo (Infections and infestations) | 2 (2)
Urethritis (Infections and infestations) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Immunisation reaction (Injury, poisoning and procedural complications) | 2 (3)
Acne (Skin and subcutaneous tissue disorders) | 2 (2)
Influenza like illness (General disorders) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT03682848/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT03682848/SAP_002.pdf